CLINICAL TRIAL: NCT00926133
Title: Impaired Glucose Tolerance in Patients With Acute Myocardial Infarction.
Brief Title: Type 2 Diabetes and Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Geir Oystein Andersen, Ullevaal University Hospital
Other Study IDs: HSØ-123
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Myocardial Infarction; Type 2 Diabetes; Impaired Glucose Tolerance; Inflammation
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus, Type 2; Glucose Intolerance; Inflammation | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples (serum,plasma) including PaxGene tubes for mRNA sampling
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI patients: Patients with acute STEMI treated by PCI without previously known type 2 diabetes.
  Interventions: Other: OGTT

INTERVENTIONS:
Other: OGTT — Oral glucose tolerance test (diagnostic procedure) eary after an acute STEMI and at three months follow-up.

SUMMARY:
The present study was designed to determine the prevalence of previously unknown impaired glucose tolerance and type 2 diabetes in patients with acute ST-elevation myocardial infarction subjected to acute PCI. Secondary, a possible association between inflammation, haemostasis and abnormal glucose regulation was studied.

DETAILED DESCRIPTION:
Background: A high prevalence of impaired glucose tolerance (IGT) and unknown diabetes mellitus (DM) in patients with cardiovascular disease has been shown. European guidelines recommend screening of patients with AMI for DM and IGT by performing an oral glucose tolerance test (OGTT). The prevalence of IGT and DM in a Norwegian population of patients with AMI is unknown. Evidence are lacking regarding the reliability of an OGTT performed early after an AMI. The present study was designed to detect unknown IGT and DM in patients with AMI and the main challenge of the study was timing and reproducibility of the OGTT. In addition, mechanisms (inflammation, haemostasis) involved in impaired glucose regulation will be studied. Design: The study is designed as an observational cohort study prospectively including 200 patients with a primary PCI treated acute STEMI admitted to the coronary care unit at Ullevål university hospital. An OGTT is performed in-hospital and repeated after 3 months and a glucometabolic classification was performed according to the results. The patients will be followed for a minimum of two-years with regards to clinical endpoints.

Aims of the study:

1. Study the prevalence of IGT and DM in a Norwegian population with acute STEMI.
2. Validate the results of an OGTT performed early after myocardial infarction, by repeating the test after three months.
3. Elucidate possible interactions between biomarkers of inflammation and coagulation, and the glucometabolic status.
4. Study the relationship between impaired glucose tolerance and prognosis after STEMI.
5. Contribute to an increased focus on undiagnosed DM and IGT in patients with coronary heart disease in Norway and the results may lead to an increased use of routine OGTT in the follow-up of patients with myocardial infarction. Investigate how patients with myocardial infarction and known glucometabolic state are followed up "in real-life" by their physicians.

Clinical implications: The study may detect a large proportion of undetected DM and IGT in patients with AMI and change present guidelines on the follow-up of patients after AMI with increased focus on impaired glucose tolerance. The study will provide new insights about the association between inflammation, haemostasis and impaired glucose tolerance in patients with acute ST-elevation myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute ST-segment elevation infarction (defined from ECG), treated with primary percutaneous coronary intervention PCI)were prospectively included.
* Stable patients

Exclusion Criteria:

* known DM
* unstable patient
* signs of heart failure
* renal failure defined as creatinine >200 umol/l

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ST-elevation myocardial infarction without known type 2-diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2005-11; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of abnormal glucose regulation defined by an oral glucose tolerance test (OGTT). | Three-months after an acute ST-elevation myocardial infarction (STEMI).

SECONDARY OUTCOMES:
Validate the results of an OGTT performed early after myocardial infarction, | Repeating the test after three months.
Elucidate possible interactions between biomarkers of inflammation and haemostasis, and the glucometabolic status. | Three months
Study the relationship between abnormal glucose regulation and prognosis after STEMI. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Geir O Andersen, MD, PhD, Study Chair — Ullevaal University Hospital; Eva C Knudsen, MD, Principal Investigator — Ullevaal University Hospital
Locations (1):
- Oslo University Hospital Ulleval, Oslo, Norway

REFERENCES:
- [Result] Knudsen EC, Seljeflot I, Abdelnoor M, Eritsland J, Mangschau A, Arnesen H, Andersen GO. Abnormal glucose regulation in patients with acute ST- elevation myocardial infarction-a cohort study on 224 patients. Cardiovasc Diabetol. 2009 Jan 30;8:6. doi: 10.1186/1475-2840-8-6. PMID 19183453
- [Derived] Helseth R, Knudsen EC, Eritsland J, Opstad TB, Arnesen H, Andersen GO, Seljeflot I. Glucose associated NETosis in patients with ST-elevation myocardial infarction: an observational study. BMC Cardiovasc Disord. 2019 Oct 15;19(1):221. doi: 10.1186/s12872-019-1205-1. PMID 31615411
- [Derived] Knudsen EC, Seljeflot I, Abdelnoor M, Eritsland J, Mangschau A, Muller C, Arnesen H, Andersen GO. Impact of newly diagnosed abnormal glucose regulation on long-term prognosis in low risk patients with ST-elevation myocardial infarction: A follow-up study. BMC Endocr Disord. 2011 Jul 29;11:14. doi: 10.1186/1472-6823-11-14. PMID 21801387
- [Derived] Knudsen EC, Seljeflot I, Abdelnoor M, Eritsland J, Mangschau A, Muller C, Arnesen H, Andersen GO. Elevated levels of PAI-1 activity and t-PA antigen are associated with newly diagnosed abnormal glucose regulation in patients with ST-elevation myocardial infarction. J Thromb Haemost. 2011 Aug;9(8):1468-74. doi: 10.1111/j.1538-7836.2011.04377.x. PMID 21624046